CLINICAL TRIAL: NCT06142149
Title: Ultrasound Versus Palpation to Find Optimal Endotracheal Tube Cuff Position in Pediatric Patients Receiving Head and Neck Surgery: Randomized Controlled Trial
Brief Title: The Optimal Endotracheal Tube Cuff Position in Pediatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun-hee Kim, Clinical associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2308-112-1459
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound group (Experimental): Use ultrasound to check the position of the endotracheal tube cuff, check its movement according to the surgical position, and position the cuff according to the size of the endotracheal tube.
  Interventions: Procedure: ultrasonographic evaluation
- Conventional group (No Intervention): Adjust the position of the endotracheal tube to account for movement in the surgical position and confirm that the endotracheal tube air sac is palpable at the suprasternal notch in the final position for surgery.

INTERVENTIONS:
Procedure: ultrasonographic evaluation — Screen the front of neck using ultrasound
  Arms: Ultrasound group

SUMMARY:
A. The hypothesis of this study is "Airway ultrasound will be superior to the conventional methods of auscultation and palpation in confirming proper positioning of the endotracheal tube in children undergoing endotracheal intubation with an endotracheal tube with cuff".

B. The purpose of this study is to determine the utility of airway ultrasound in confirming proper positioning of the endotracheal tube.

C. In addition, we would like to suggest what criteria should be used when using airway ultrasound to determine the fixed position of an endotracheal tube.

DETAILED DESCRIPTION:
1. Obtain consent from the guardian of the target patient before surgery and perform randomization.
2. After entering the operating room, attach equipment for electrocardiogram, non-invasive blood pressure, peripheral oxygen saturation, anesthesia depth monitoring, and neuromuscular blockade monitoring.
3. Prepare the endotracheal tube according to the patient's age. 6 months to 18 months: internal diameter 3.5 18 months to 2 years: internal diameter 3.5 or 4.0 2-4 years: internal diameter 4.0 4 to 5 years: internal diameter 4.5 5 years and older: Age/4 + 3.5
4. When sufficient neuromuscular blockade is achieved after infusion of neuromuscular blocking agents, after inserting the endotracheal tube, check the position of the endotracheal tube according to the assigned group, fix the endotracheal tube in consideration of changes in posture during surgery, and record its depth.

   Ultrasound group A. During tracheal intubation using a video laryngoscope, the endotracheal tube is stopped when the endotracheal tube cuff passes through the vocal cord.

   B. Use ultrasound to check the position of the endotracheal tube cuff, check its movement according to the surgical position, and position the cuff according to the size of the endotracheal tube as follows.
   * internal diameter 3.5, internal diameter 4.0: The cuff is positioned 0.5 cm below the lower margin of the cricoid cartilage.
   * internal diameter 4.5, internal diameter 5.0: The cuff is positioned 1 cm below the lower margin of the cricoid cartilage.

   C. In the final position, check for bilateral lung movement (lung sliding sign) using lung ultrasound.

   D. Record the depth of fixation of the endotracheal tube.

   Conventional Group A. During tracheal intubation with video laryngoscope, stop the endotracheal tube when the cuff of the endotracheal tube passes through the vocal cords, and confirm that the cuff of the endotracheal tube is palpable at the suprasternal notch.

   B. Adjust the position of the endotracheal tube to account for movement in the surgical position and confirm that the endotracheal tube cuff is palpable at the suprasternal notch in the final position for surgery.

   C. Confirm that bilateral lung sounds are audible through auscultation and secure the endotracheal tube.

   D. Record the depth of endotracheal tube placement.
5. After the end of surgery and before awakening the patient, check the position of the endotracheal tube cuff using ultrasound.

Record how far the proximal margin of the endotracheal tube cuff is from the lower margin of the cricoid and how it relates to surrounding structures (1st tracheal ring, 2nd tracheal ring, 3rd tracheal ring, below the 3rd tracheal ring, above the cricoid level).

Check the movement of both lungs (sliding sign) using lung ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients ages 6 months to 7 years who are scheduled to have an endotracheal tube inserted for facial or intraoral surgery.

Exclusion Criteria:

* When difficult intubation is anticipated
* If the patient has deformities such as facial asymmetry due to congenital causes such as genetic diseases or acquired causes such as accidents.
* If the patient or guardian does not agree to participate in the study.
* Other cases deemed unsuitable by the researcher

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
percentage of the patients whose cuff is optimally located. | at the end of the surgery
  Percentage of patients with endotracheal tube cuff located below the cricoid lower margin and at a depth that allows movement of both lungs, as confirmed by postoperative ultrasound.

SECONDARY OUTCOMES:
Differences in final endotracheal tube fixation depth in the two groups | at the end of induction of anesthesia
  difference between tube fixation depth (cm)
Incidence of respiratory events | throughout the surgery
  endobronchial intubation, incidental extubation, laryngospasm, bronchospasm, desaturation, airway obstruction, stridor
proportion of final cuff position | at the end of the surgery
  Above cricoid / 1st ring / 2nd ring / 3rd ring / below 3rd ring of trachea
incidence of postoperative complication | at postanesthetic care unit
  laryngospasm, bronchospasm, desaturation, airway obstruction, stridor, severe coughing

CONTACTS AND LOCATIONS:
Overall Officials: Eun-Hee Kim, M.D., Ph.D., Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Limited availability to those deemed appropriate by the researcher.